CLINICAL TRIAL: NCT00750841
Title: A Phase I, Open Label, Non-Randomised Study to Assess the Effect of Rifampicin on the Pharmacokinetics of Multiple Oral Doses of Cediranib (AZD2171, RECENTIN™), in Patients With Advanced Solid Tumours
Brief Title: Study of the Effect of Rifampicin on the Pharmacokinetics (PK) of Multiple Doses of Cediranib in Patients With Solid Tumours
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D8480C00029; 2008-002519-42 (EudraCT Number)
Record Dates: First submitted 2008-09-10; First posted 2008-09-11 (Estimated); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Solid Tumors
Keywords: advanced cancer; metastatic; rifampicin; pharmacokinetics; Phase I; Advanced solid tumours
MeSH Terms: conditions — Neoplasm Metastasis | interventions — cediranib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Cediranib alone, followed by cediranib plus rifampicin, followed by cediranib alone.
  Interventions: Drug: cediranib

INTERVENTIONS:
Drug: cediranib — 45 mg cediranib once daily from Days 1-7; cediranib 45 mg plus 600 mg rifampicin from Days 8-14; 45 mg cediranib once daily from Days 15-28; from Day 29 patients may continue on 45 mg cediranib or dose reduce.
  Other Names: RECENTIN

SUMMARY:
Phase I, open study to assess the effect of rifampicin, a marketed drug, on how the body handles the experimental drug cediranib in patients with advanced cancer.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Prostate cancer), which is refractory to standard therapies or for which no standard therapy exists.
* Estimated life expectancy of at least 8 weeks
* WHO performance status (PS) 0-2.

Exclusion Criteria:

* Unstable brain/meningeal metastases
* Biochemistry/haematology results outside of required ranges
* History of significant GI impairment
* Inadequate bone marrow reserve

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2008-09-09 (Actual); Primary Completion 2009-07-30 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
To assess the steady-state PK parameters of cediranib in the presence and absence of rifampicin | PK assessments to be taken until Day 28. Days 7 and 14 PK parameters used to assess the primary variables.

SECONDARY OUTCOMES:
To assess the safety and tolerability of cediranib in the presence of rifampicin, by assessment of Adverse events (AEs) Laboratory findings, Vital signs, physical examination and Electrocardiogram. | Until study drug is discountinued

CONTACTS AND LOCATIONS:
Overall Officials: Michael Sawyer, MD, Principal Investigator — Cross Cancer Institute, Edmonton, AB, Canada
Locations (5):
- Canada (2):
  - Research Site, Edmonton, Alberta
  - Research Site, Montreal, Quebec
- United Kingdom (3):
  - Research Site, Dundee
  - Research Site, Glasgow
  - Research Site, London

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: CSR-D8480C00029.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=628&filename=CSR-D8480C00029.pdf